CLINICAL TRIAL: NCT00088972
Title: Randomized Placebo-Controlled Biomarker Modulation Trial Using Celecoxib in Premenopausal Women at High Risk for Breast Cancer
Brief Title: S0300, Celecoxib in Preventing Breast Cancer in Premenopausal Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to poor accrual.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000377698; U10CA012027 (NIH); S0300 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast cancer in situ; lobular breast carcinoma in situ; ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Ductal, Breast | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I - Celecoxib (Experimental): Patients receive oral celecoxib twice daily for 12 months in the absence of unacceptable toxicity or diagnosis of cancer.
  Interventions: Drug: celecoxib
- Arm II - Placebo (Placebo Comparator): Patients receive oral placebo twice daily for 12 months in the absence of unacceptable toxicity or diagnosis of cancer.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: celecoxib — Given orally
  Arms: Arm I - Celecoxib
Other: placebo — Given orally
  Arms: Arm II - Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of celecoxib may be effective in preventing breast cancer.

PURPOSE: This randomized phase II trial is studying how well celecoxib works in preventing breast cancer in premenopausal women who are at risk for developing the disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare 1-year mammographic density in premenopausal women at high risk for developing breast cancer treated with celecoxib vs placebo.
* Compare 1-year proliferation of breast epithelial cells, as measured by Ki67 staining, in patients treated with these drugs.
* Compare the expression of other biomarkers, including cyclo-oxygenase-2 (COX-2) enzyme and a marker of apoptosis, in breast tissue of patients treated with these drugs.
* Compare 1-year plasma levels of insulin-like growth factor (IGF)-1, IGF binding protein-3, and prostaglandin E_2 in patients treated with these drugs.
* Compare the toxicity of these drugs in these patients.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to risk category (lobular carcinoma in situ or ductal carcinoma in situ vs BRCA1/2 mutation AND any Gail risk vs Gail risk ≥1.7% but < 5% vs Gail risk ≥ 5%) and prior tamoxifen use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Celocoxib: Patients receive oral celecoxib twice daily.
* Placebo: Patients receive oral placebo twice daily. In both arms, treatment continues for 12 months in the absence of unacceptable toxicity or diagnosis of cancer.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At elevated risk of developing breast cancer, as defined by 1 of the following:

  * Modified Gail risk at 5 years ≥ 1.7% or lifetime risk ≥ 20% AND Claus Model, BRCAPro Model, or Tyrer-Cuzick Model lifetime risk ≥ 20%
  * Diagnosis of lobular carcinoma in situ or ductal carcinoma in situ
  * Known deleterious mutation of BRCA1 or BRCA2
* At least 1 breast available for imagery and biopsy
* Has undergone a baseline mammogram with a standard density wedge within 7-14 days after completion of the last menstrual period AND within 7 days before study entry

  * Mammogram normal or benign (BIRADS score 0 or 1)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Premenopausal, defined by 1 of the following criteria:

  * Last menstrual period < 6 months ago AND no prior bilateral ovariectomy AND not on estrogen replacement therapy
  * Prior hysterectomy (with ovaries still in place) AND normal follicle-stimulating hormone levels within 28 days of study entry

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2.0 times institutional upper limit of normal (IULN)
* SGOT or SGPT < 2 times IULN
* Alkaline phosphatase < 2 times IULN
* INR ≤ 1.5
* PT and PTT ≤ IULN

Renal

* Serum creatinine < 2.0 times IULN

Cardiovascular

* No history of myocardial infarction
* No angina pectoris
* No known coronary artery disease
* No history of stroke or mini-stroke (e.g., transient ischemic attack)
* No history of thromboembolic disease (e.g., deep vein thrombosis or pulmonary embolism)
* No uncontrolled hypertension (i.e., blood pressure > 140/90 mmHg)

Pulmonary

* No asthma after taking aspirin or other NSAIDs

Other

* No known sensitivity to celecoxib
* No allergy to sulfonamides
* No urticaria or allergic-type reactions after taking aspirin or other NSAIDs
* No extreme lactose intolerance
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or early bladder cancer (preinvasive transitional cell carcinoma of the bladder)
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 5 years since prior biologic therapy for cancer

Chemotherapy

* More than 5 years since prior chemotherapy for cancer

Endocrine therapy

* At least 28 days since prior tamoxifen
* No prior systemic estrogen modifiers (SERMs) or aromatase inhibitors
* Concurrent hormonal contraception (i.e., pills, patches, or shots) allowed provided contraception was initiated prior to study entry

Radiotherapy

* No prior radiotherapy to the breast to be studied

Surgery

* Not specified

Other

* At least 7 days since prior anticoagulant therapy
* More than 1 month since prior chronic daily aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) of more than 7 days duration

  * Concurrent intermittent aspirin or NSAIDs allowed (no more than 10 days per month)
* No concurrent participation in another clinical trial for treatment or prevention of cancer unless no longer receiving treatment and is in the follow-up phase

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Powel H. Brown, MD, PhD, Study Chair — Baylor College of Medicine
Locations (9):
- United States (9):
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive oral celecoxib twice daily for 12 months in the absence of unacceptable toxicity or diagnosis of cancer.
- Arm II: Patients receive oral placebo twice daily for 12 months in the absence of unacceptable toxicity or diagnosis of cancer.
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 3 | 5
Completed | 1 | 1
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (3.9) | 43.3 (5.9) | 43.5 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mammographic Density
Description: The primary outcome measure is change in mammographic density. The null hypothesis is that there is no difference between the arms in change in mammographic density over one year versus the alternative that the treatment arm reduces mammographic density by 10 points (percent of pixels highlighted) or more over one year compared to the change in the placebo arm.
Time Frame: 1 year
Population: Counts represent number of patients for by arm for whom a 1 year mammographic density image was submitted. However, since the study was closed early due to poor accrual, there was insufficient accrual to evaluate study endpoints, and these images were never analyzed.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Ki-67 Expression
Description: The difference between the two arms in the percent of patients with non-zero ki-67 expression over the two time periods (baseline and 1-year).
Time Frame: 1 year
Population: Since the study was closed early due to insufficient accrual, the ki-67 data were never collected.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=3) | Arm II (N=5)
Pain - breast (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Grade 1
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) — Grade 1
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No